CLINICAL TRIAL: NCT02921074
Title: STATE Trial: SusTained Attention Training to Enhance Sleep
Acronym: STATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1009-16
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Experimental Treatment (Experimental): Computerized plasticity-based adaptive cognitive training requiring a total maximum of 24 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training
- Active Comparator (Active Comparator): Commercially available computerized training requiring a total maximum of 24 treatment sessions, up to 7 sessions per week, 36 minutes per session.
  Interventions: Other: Commercially available computerized training

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training
  Arms: Experimental Treatment
Other: Commercially available computerized training
  Arms: Active Comparator

SUMMARY:
This study is a validation study to document the acceptability of the Tonic and Phasic Alertness Training (TAPAT) training program in older adults with chronic late-life insomnia. The goal of this study is to employ a computerized attention-training program, TAPAT, designed for chronic late-life insomnia in a randomized, controlled trial to assess feasibility and initial efficacy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be between ages 55 and 80.
* Participant must meet current diagnostic criteria for Primary Insomnia Disorder based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5).
* Participant with hypertension must be undergoing treatment for this condition and on a stable medication regimen for hypertension for ≥ 8 weeks prior to screening.
* Participant must be a fluent English speaker
* Participant must have adequate visual, auditory, and motor capacity to use computerized intervention
* Participant must be willing to wear Microsoft Band 2 watch to track sleep patterns

Exclusion Criteria:

* Participants with cognitive impairment, delirium or dementia, or evidence of cognitive impairment from a pre-existing cause.
* Participants with untreated psychiatric conditions, including substance abuse/dependence disorders, untreated obstructive sleep apnea, diagnosis of other sleep disorders (e.g., restless legs syndrome), recent hospitalization, ongoing chemotherapy or other cancer treatment, and concurrent engagement in another insomnia treatment.
* Participants enrolled in another concurrent research study.
* Participants who have difficulty performing assessments or comprehending or following spoken instructions, in the judgment of the screening clinician.
* Participants using computer-based cognitive training programs or has used them within a month of the consent date.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-10 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency and sleep duration scores on the Pittsburg Sleep Quality Index | 4 months
Sleep duration obtained by actigraphy (Microsoft Band 2 watch) | 4 months
Sleep duration obtained by sleep diary | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Posit Science Corporation, San Francisco, California, United States